CLINICAL TRIAL: NCT07235150
Title: A PHASE 1, RANDOMIZED, MULTI-CENTER, DOUBLE-BLIND, SPONSOR OPEN, PLACEBO-CONTROLLED, SINGLE DOSE-ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF PF-07985631 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-07985631 Are Tolerated and Act in the Body in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C5661003
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: healthy participants; healthy volunteers; safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort 1 Dose A (3 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be subcutaneous (SC)
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 2 Dose B (3 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 3 Dose C (6 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 4 Dose D (6 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 5 Dose E (6 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 6 Dose F (6 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 7 Dose G (6 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 8 Optional Cohort with dose to be determined, Japanese (4 active: 1 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 9 Optional Cohort with dose to be determined, Chinese (4 active: 1 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 10 Optional Cohort with dose to be determined (6 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo
- Cohort 11 Optional Cohort with dose to be determined (6 active: 2 placebo) (Experimental): Drug: PF-07985631 Experimental Pfizer compound which will be SC
  Drug: Placebo Placebo which will be SC
  Interventions: Drug: PF-07985631; Drug: Placebo

INTERVENTIONS:
Drug: PF-07985631 — Experimental Pfizer compound which will be SC
Drug: Placebo — Placebo which will be SC

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called PF-07985631) for the possible treatment of a kidney disease called IgA nephropathy.

This study is seeking participants who

* are male or female between 18 and 45 years of age (55 for Japanese/Chinese/multiple dose participants)
* are deemed to be healthy Participants in this study will receive PF-07985631 or placebo. A placebo does not have any medicine in it but looks just like the medicine being studied.

PF-07985631 or placebo will be given as a small needle injection (in the abdomen, thigh or back of the arm) at the study clinic. Most participants will receive PF-07985631 or placebo one time. Some participants may receive PF-07985631 or placebo twice.

The study will compare the experiences of people receiving PF-07985631 to those of the people who do not. This will help decide if PF-07985631 is safe and effective.

Participants who take PF-07985631 or placebo will take part in this study for about four- four and a half months. During this time, they will stay at the study clinic for 12 to 19 days and will have 7 more study visits at the study clinic.

During study clinic stays and study visits, blood samples will be done and safety reviews completed.

ELIGIBILITY:
Inclusion:

1. Between 18 and 45 years of age who are overtly healthy.
2. Japanese/Chinese cohorts only: Adult participants 18 to 55 years of age
3. Japanese/Chinese cohorts only: Participants must have 4 biological Japanese/Chinese grandparents who were born in Japan/China.

Exclusion:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Participants with a history of allergic or anaphylactic reaction with any investigative biologic agents.
3. History of infections requiring treatment within 28 days prior to Day 1 or any active infection at Day 1.
4. Active or latent infection with tuberculosis.
5. History of recurrent urinary tract infections AND/OR sinopulmonary infections AND/OR gastrointestinal infections requiring antibiotic treatment.
6. Known fever within the 7 days prior to dosing.
7. Active gastrointestinal (GI) tract ulcerations or GI bleeding.
8. Vaccination within 6 weeks prior to Day 1 dosing or planned vaccination during the study.
9. Positive urine drug test.
10. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic).
11. Estimated glomerular filtration rate (eGFR) <75 mL/min/1.73 m².
12. Chest X-ray showing any active disease in the chest, or pulmonary nodules >0.5 cm in diameter that have not been previously evaluated, cavitary lesions or evidence of bronchiectasis.
13. Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
14. Positive stool hematest at screening or admission.
15. Participants with ANY of the following abnormalities in clinical laboratory tests at screening:

    * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (direct and total) ≥1.05 × upper limit of normal
    * Immunoglobulin G, Immunoglobulin M, Immunoglobulin A below the lower limit of normal (LLN)
    * Total white blood cell (WBC) below the LLN
    * Lymphocyte count below the LLN
    * Platelet count below the LLN
    * Hemoglobin below the LLN

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-07-27 (Estimated); Study Completion 2027-07-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAE) | Baseline (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)
Number of Participants With Clinically Significant Abnormal Laboratory Parameters | Baseline (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)
Number of Participants With Vital Signs Values Meeting Categorical Summarization Criteria | Baseline (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)
Number of Participants With Notable Electrocardiogram (ECG) Values | Baseline (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) as data permit | Predose (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) as data permit | Predose (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)
Maximum Observed Plasma Concentration (Cmax) as data permit | Predose (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)
Time to Reach Maximum Observed Plasma Concentration (Tmax) as data permit | Predose (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)
Plasma Decay Half-Life (t1/2) as data permit | Predose (Day 1) up to 83 days after last dose of study drug (approximately up to 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Q-Pharm Pty Ltd. (Nucleus Network), Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5661003